CLINICAL TRIAL: NCT01138371
Title: Inflammatory and Lipid Markers Pre- and Post-LDL Apheresis: A Multicenter Experience
Brief Title: Effects of Low-density Lipoprotein (LDL) Apheresis on Inflammatory and Lipid Markers
Acronym: INFLAME
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: Kaneka Medical America LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB00044778; INFLAME_EUH (Other: Other)
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Familial Hypercholesterolemia
Keywords: LDL apheresis; Familial hypercholesterolemia; Inflammatory markers; Hyperlipidemia; Cardiovascular disease
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Hyperlipidemias; Cardiovascular Diseases | interventions — Blood Component Removal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples only
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Familial hypercholesterolemia: * Heterozygous FH with documented CAD and LDL-C ≥ 200 mg/dL (Documented CAD may be represented as: Lesion(s) on coronary angiography, history of myocardial infarction, CABG, PTCA, progressive angina demonstrated by stress testing, history of other revascularization procedure)
  * Homozygous FH and LDL-C > 500 mg/dL
  * Heterozygous FH and LDL-C ≥ 300 mg/dL
  * On stable LDL apheresis therapy for at least 6 months
  Interventions: Procedure: LDL Apheresis

INTERVENTIONS:
Procedure: LDL Apheresis — LDL Apheresis
  Other Names: Apheresis; LDL filtration

SUMMARY:
The primary objective of this study is to measure how LDL apheresis affects levels of inflammatory and cholesterol markers in human beings. The investigators will address this question by drawing pre- and post-LDL apheresis blood from patients who are undergoing this procedure. A secondary objective of this study is to learn how specific inflammatory markers behave in our blood in terms of time to rebound back to normal levels. The investigators will address this question by drawing post-LDL apheresis blood at predetermined time intervals.

DETAILED DESCRIPTION:
Numerous epidemiological investigations have demonstrated the importance of cholesterol - specifically low density lipoprotein (LDL) - in the development and progression of atherosclerosis. A continuing relationship between cholesterol level and coronary morbidity has been established. The initial approach for managing elevated cholesterol includes lifestyle interventions, namely eating a low fat diet, weight loss in overweight patients, and regular aerobic exercise. Once lifestyle interventions have been applied, pharmacologic therapy becomes a mainstay of therapy, conventionally with a statin followed by adjunctive medicines as indicated. Certain populations that are refractory to aggressive pharmacotherapy, however - such as patients who have familial hypercholesterolemia (FH) - necessitate alternative means of lipid management. Therapeutic considerations in these patients include LDL apheresis and a number of rare procedures such as partial ileal bypass, liver transplantation, portocaval shunting, and possibly gene therapy in the future.

The anti-inflammatory effects of LDL apheresis and its effects on endothelial function are not well known. Considering several pathways of atherogenesis, and inflammation as a central mechanism thereof, LDL apheresis may theoretically provide synergistic benefit of lipid lowering as well as proinflammatory agent lowering that can lead to significantly decreased atherogenesis. This study looks to address these questions by assessing the effects of LDL apheresis on inflammatory and lipid markers.

ELIGIBILITY:
Inclusion criteria:

* Heterozygous FH with documented CAD and LDL-C ≥ 200 mg/dL Documented CAD may be represented as: Lesion(s) on coronary angiography, history of myocardial infarction, CABG, PTCA, progressive angina demonstrated by stress testing, history of other revascularization procedure (e.g. atherectomy)
* Homozygous FH and LDL-C > 500 mg/dL
* Heterozygous FH and LDL-C ≥ 300 mg/dL
* On stable LDL apheresis therapy for at least 6 months.

Exclusion criteria:

* Patient refusal to participate
* Inability to attend 2 consecutive LDL apheresis sessions for study duration
* Subject with advanced renal disease
* Subject with chronic progressive hepatic disease and demonstrated deficient synthetic function
* Subject with acute hepatic process
* Subject with current malignancy
* Subject with diagnosis of amyloidosis
* Subject with diagnosis of rheumatoid arthritis
* Any subject with acute flare of chronic disease
* Subject with recent ethanol ingestion
* Subject with significant bone disease

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study focuses on people who are currently on stable LDL apheresis treatment for high cholesterol.
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2011-03; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Lipid Marker Change | 1 month
  We will measure the level of cholesterol markers in your blood before and after the LDL apheresis procedure with a blood draw.
Inflammatory Marker Change | 1 month
  We will measure the level of inflammatory markers in your blood before and after the LDL apheresis procedure with blood draws (for 2 apheresis sessions)

SECONDARY OUTCOMES:
Inflammatory Marker Rebound | 2 days
  We will measure the level of inflammatory markers in your blood after LDL apheresis procedure the following morning, 24 hours after procedure, and on the second morning.

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Sperling, MD, Principal Investigator — Emory University; Vimal Ramjee, MD, Study Director — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Background] Napoli C, Ambrosio G, Scarpato N, Corso G, Palumbo G, D'Armiento FP, Mancini FP, Malorni A, Formisano S, Ruocco A, Cali A, Chiariello M. Decreased low-density lipoprotein oxidation after repeated selective apheresis in homozygous familial hypercholesterolemia. Am Heart J. 1997 May;133(5):585-95. doi: 10.1016/s0002-8703(97)70155-8. PMID 9141382
- [Background] Mehta PK, Baer J, Nell C, Sperling LS. Low-density lipoprotein apheresis as a treatment option for hyperlipidemia. Curr Treat Options Cardiovasc Med. 2009 Aug;11(4):279-88. doi: 10.1007/s11936-009-0029-1. PMID 19627661
- [Background] Mabuchi H, Higashikata T, Kawashiri MA. Clinical applications of long-term LDL-apheresis on and beyond refractory hypercholesterolemia. Transfus Apher Sci. 2004 Jun;30(3):233-43. doi: 10.1016/j.transci.2004.01.006. PMID 15172629
- [Background] Thompson GR. LDL apheresis. Atherosclerosis. 2003 Mar;167(1):1-13. doi: 10.1016/s0021-9150(02)00251-4. PMID 12618263
- [Background] Thompson GR, Maher VM, Matthews S, Kitano Y, Neuwirth C, Shortt MB, Davies G, Rees A, Mir A, Prescott RJ, et al. Familial Hypercholesterolaemia Regression Study: a randomised trial of low-density-lipoprotein apheresis. Lancet. 1995 Apr 1;345(8953):811-6. doi: 10.1016/s0140-6736(95)92961-4. PMID 7898227
- [Background] Kroon AA, Aengevaeren WR, van der Werf T, Uijen GJ, Reiber JH, Bruschke AV, Stalenhoef AF. LDL-Apheresis Atherosclerosis Regression Study (LAARS). Effect of aggressive versus conventional lipid lowering treatment on coronary atherosclerosis. Circulation. 1996 May 15;93(10):1826-35. doi: 10.1161/01.cir.93.10.1826. PMID 8635262
- [Background] Igarashi K, Tsuji M, Nishimura M, Horimoto M. Improvement of endothelium-dependent coronary vasodilation after a single LDL apheresis in patients with hypercholesterolemia. J Clin Apher. 2004;19(1):11-6. doi: 10.1002/jca.20000. PMID 15095396
- [Background] Tamai O, Matsuoka H, Itabe H, Wada Y, Kohno K, Imaizumi T. Single LDL apheresis improves endothelium-dependent vasodilatation in hypercholesterolemic humans. Circulation. 1997 Jan 7;95(1):76-82. doi: 10.1161/01.cir.95.1.76. PMID 8994420
- [Background] Kobayashi S, Moriya H, Maesato K, Okamoto K, Ohtake T. LDL-apheresis improves peripheral arterial occlusive disease with an implication for anti-inflammatory effects. J Clin Apher. 2005 Dec;20(4):239-43. doi: 10.1002/jca.20033. PMID 15880405
- [Background] Moriarty PM, Gibson CA. Effect of low-density lipoprotein apheresis on lipoprotein-associated phospholipase A2. Am J Cardiol. 2005 May 15;95(10):1246-7. doi: 10.1016/j.amjcard.2005.01.058. PMID 15878003
- [Background] Wang Y, Blessing F, Walli AK, Uberfuhr P, Fraunberger P, Seidel D. Effects of heparin-mediated extracorporeal low-density lipoprotein precipitation beyond lowering proatherogenic lipoproteins--reduction of circulating proinflammatory and procoagulatory markers. Atherosclerosis. 2004 Jul;175(1):145-50. doi: 10.1016/j.atherosclerosis.2004.03.011. PMID 15186959
- [Background] Nakamura T, Matsuda T, Suzuki Y, Ueda Y, Koide H. Effects of low-density lipoprotein apheresis on plasma matrix metalloproteinase-9 and serum tissue inhibitor of metalloproteinase-1 levels in diabetic hemodialysis patients with arteriosclerosis obliterans. ASAIO J. 2003 Jul-Aug;49(4):430-4. PMID 12918586
- [Background] Hovland A, Hardersen R, Sexton J, Mollnes TE, Lappegard KT. Different inflammatory responses induced by three LDL-lowering apheresis columns. J Clin Apher. 2009;24(6):247-53. doi: 10.1002/jca.20223. PMID 19927364
- [Background] Kojima S, Shida M, Yokoyama H. Changes in C-reactive protein plasma levels during low-density lipoprotein apheresis. Ther Apher Dial. 2003 Aug;7(4):431-4. doi: 10.1046/j.1526-0968.2003.00080.x. PMID 12887727